CLINICAL TRIAL: NCT07187895
Title: Comparative Imaging Study of PET Myocardial Perfusion With XTR004 Injection Versus MIBI SPECT in Patients With Borderline Coronary Stenosis
Brief Title: Comparative Imaging of XTR004 PET and MIBI SPECT in Borderline Coronary Stenosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The main objective of this study has been achieved. Following internal discussions, the sponsor has decided to terminate this study early.
Sponsor: Sinotau Pharmaceutical Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STB-XTR004-202
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Myocardial Perfusion Imaging; Diagnostic Certainty; Stable Coronary Artery Disease
Keywords: XTR004; MPI; PET; SPECT; diagnostic certainty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XTR004 MPI PET & MIBI SPECT MPI (Experimental): Patients with suspected or known stable coronary artery disease who have previously undergone coronary CTA showing 30%-80% stenosis in any coronary vessel, or mild to moderate stenosis, will be enrolled and sequentially undergo MIBI SPECT myocardial perfusion imaging (MPI) and XTR004 PET MPI
  Interventions: Drug: XTR004

INTERVENTIONS:
Drug: XTR004 — At rest: IV bolus injection of XTR004 with a dose range of 2.0-2.5 mCi
  At stress: IV infusion of adenosine at a rate of 140 μg/kg/min. IV bolus injection of XTR004 with a dose range of 6.0-7.5 mCi.

SUMMARY:
Compare the diagnostic certainty of MIBI SPECT myocardial perfusion imaging (MPI) and XTR004 PET MPI.

DETAILED DESCRIPTION:
This trial is a single-arm, single-center, open-label, self-controlled study. Patients with suspected or known stable coronary artery disease who have previously undergone coronary CTA showing 30%-80% stenosis in any coronary vessel, or mild to moderate stenosis, will be enrolled and sequentially undergo MIBI SPECT myocardial perfusion imaging (MPI) and XTR004 PET MPI. Imaging will be independently and blindly read by expert readers for both MIBI SPECT MPI and XTR004 PET MPI. The diagnostic certainty of the reading results from the two imaging modalities will then be compared.

ELIGIBILITY:
Inclusion Criteria:

* 1.Male or female participants aged 18 years or older.
* 2.Suspected or known stable coronary artery disease with related symptoms and stable condition, and having at least one coronary artery disease risk factor, including: hypertension, hyperlipidemia, diabetes, obesity, alcohol abuse, smoking, family history of coronary artery disease, postmenopausal status in women, or advanced age.
* 3.Underwent coronary CTA within the past 6 months showing 30%-90% stenosis, or indicating mild to moderate-to-severe stenosis.
* 4.Able to communicate effectively with the investigators, understand and comply with the clinical study requirements, voluntarily participate in the study, and provide written informed consent.

Exclusion Criteria:

* 1. Patients with a history of percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG).
* 2.Patients with a prior diagnosis of myocardial infarction, congenital heart disease, cardiomyopathy, myocarditis, or other cardiac diseases.
* 3.Patients known to have severe allergic reactions to alcohol.
* 4.Patients known to have an allergy or other contraindications to adenosine.
* 5.Patients known to be allergic to iodinated contrast agents.
* 6.Individuals with significant occupational exposure to ionizing radiation within the past 10 years (e.g., exceeding 50 mSv/year), or exposure to radioactive substances or ionizing radiation for therapeutic or research purposes.
* 7.Men and women of childbearing potential who do not plan to use effective contraception during the study and for 6 months after study completion (effective methods include sterilization, intrauterine hormonal devices, condoms, contraceptive pills/agents, abstinence, or partner vasectomy/tubal ligation).
* 8.Pregnant or lactating women.
* 9.Patients with claustrophobia, bipolar disorder, other psychiatric disorders, or poor compliance.
* 10.Patients who participated in another investigational drug clinical study within 30 days prior to enrollment or plan to do so during follow-up.
* 11.Any other condition that, in the opinion of the investigators, makes the patient unsuitable for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2024-12-19 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Percentage of vessel-level diagnostic certainty for XTR004 PET/MIBI SPECT myocardial perfusion imaging. | Day1-7

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes